CLINICAL TRIAL: NCT06347536
Title: Supported Rescue Packs Post-discharge in Chronic Obstructive Pulmonary Disease: An Open-label Multicenter Randomised Controlled Trial
Brief Title: Supported Rescue Packs Post-discharge in Chronic Obstructive Pulmonary Disease
Acronym: RAPID
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other); University College, London (Other); Imperial College London (Other); University of Cambridge (Other); University of Southampton (Other); University of Nottingham (Other); University of Leicester (Other); Frimley Health NHS Foundation Trust (Unknown); Newcastle University (Other); University of Bristol (Other); Asthma and Lung UK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS331831; NIHR156698 (Other Grant/Funding Number: NIHR HTA)
Record Dates: First submitted 2024-02-19; First posted 2024-04-04 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: COPD; COPD Exacerbation
Keywords: COPD; exacerbation; hospital admission; rescue packs; self-management support
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supported Rescue Pack Arm (Experimental): All patients in the SRP arm will receive 1) a rescue pack (prednisolone and antibiotics for 5 days); 2) a written rescue pack management plan based on the Asthma-Lung UK plan; and 3) twice-weekly automated telephone symptom reminder calls for 90 days (with preferred language as needed). The reminder phone calls (to home telephone or mobile) will ask questions aligned to the written management plan, with patients asked to press the telephone keys 0-9 depending on the answer to the questions. Any patient that has required the use of their rescue pack within 90 days of discharge, will be re-issued with a rescue pack by the central study team and will be sent to the patient home.
  Interventions: Combination Product: Supported rescue pack
- No Rescue Pack Arm (No Intervention): In this arm, patients will be randomised to receive no rescue packs on discharge. We will very carefully characterise the support provided to people in this arm, upon discharge from hospital, including any access to rescue packs in the community (which we will report, but not modify).

INTERVENTIONS:
Combination Product: Supported rescue pack — 1) a rescue pack (prednisolone and antibiotics for 5 days); 2) a written rescue pack management plan based on the Asthma-Lung UK plan; and 3) twice-weekly automated telephone symptom reminder calls for 90 days (with preferred language as needed). The reminder phone calls (to home telephone or mobile) will ask questions aligned to the written management plan
  Arms: Supported Rescue Pack Arm

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic lung disease affecting approximately 10% of the adult population globally. COPD is recognised to be an important area of focus, as part of one of the healthcare challenges defined by the Office of Life Sciences. Patients with COPD often experience exacerbations which are triggered episodes leading to disease worsening. Exacerbations are associated with increased morbidity and a risk of mortality.

Severe exacerbations, where patients are hospitalised, are of particular concern to patients, carers and healthcare givers. The National Institute for Health and Care Excellence (NICE) recommends that hospital clinicians looking after patients with COPD should provide rescue packs (a course of prednisolone and antibiotics) and a basic management plan to patients on discharge. It is recognised that there is a high-risk 90-day period to patients with COPD following discharge from hospital, where there is a 43% risk of readmission and a 12% risk of mortality; however repeated national audit data has shown that, despite NICE recommendations this high risk of readmission and mortality has not changed.

A multicentre randomised clinical trial of 1400 patients will be conducted in 30 acute NHS trusts. This will test the hypothesis that a self-supported rescue pack management plan consisting of rescue packs + written self-management plan + twice weekly telephone/text symptom alert assessments in the high-risk 90-day period is better than standard care in reducing 90-day readmission by 20%. If successful, this intervention would be rapidly implementable, improve patient clinical outcomes and have a cost saving of approximately £350 million per annum.

DETAILED DESCRIPTION:
What is the problem being addressed?

Chronic obstructive pulmonary disease (COPD) is a common lung condition in the United Kingdom, with a prevalence of 4.5% in population ≥40 years and rising4. In addition to daily symptoms such as cough and breathlessness that limit physical activity, people living with COPD are prone to unpredictable deteriorations in their health called 'exacerbations'. Exacerbations are sometimes severe enough to lead to hospital admission and are often driven by infections. A systematic review of patient outcomes in COPD identified exacerbations, especially severe hospitalised exacerbations, as the aspect of COPD that patients found most difficult to live with. Prior to the pandemic there were around 115,000 admissions to hospital with COPD exacerbations per annum6 and admissions are now returning to that level. Exacerbations are more common in the winter with greater circulation of respiratory viruses, and thus the burden of hospitalised exacerbations contributes to winter National Health Service (NHS) bed pressures and cost to the NHS. The annual healthcare cost for people with moderate and severe exacerbation of COPD in England was estimated to be nearly £1 billion in 20227. A particular problem after a hospitalised COPD exacerbation is re-admission to hospital. The National Asthma and COPD Audit Programme (NACAP) has shown that the re-admission rate is 23% at 30 days and 43% at 90 days2. A systematic review conducted by the authors identified comorbidities, previous exacerbations and increased length of stay as risk factors for 30- and 90-day all-cause readmission5.

There are many interventions that can reduce the risk of COPD exacerbations but these are incompletely effective8. There is also evidence to suggest that earlier intervention with standard exacerbation treatment of antibiotics and/or corticosteroids (called a 'rescue pack') can hasten recovery, with a lessened chance of hospital admission9. As part of standard NHS care2, patients with COPD should have a 'discharge bundle' implemented, although this is often poorly delivered and has not been definitively shown to impact outcomes (likely because the wrong outcomes were chosen, and the bundle was poorly implemented)10. The provision of rescue packs is not a standard component of discharge bundles but these are sometimes provided according to local service preference3. Additionally, in usual clinical practice, some patients will have been prescribed rescue packs from primary care (GP) or a community respiratory team (CRT) prior to being hospitalised with COPD. Furthermore, patients may or may not have access to rescue packs from the GP or the CRT after hospital discharge.

Although rescue packs are part of NICE guidance2, the available evidence suggests they are not effective unless provided in the context of a more comprehensive management/education plan that supports patients in their appropriate use11. In practice this usually does not happen3, with evidence that a patient with COPD will receive variable or often no support; with some patients receiving rescue packs on demand without considering antimicrobial resistance, predictable side-effects from steroid overuse, or reviewing appropriateness. The investigators have pilot data that show receiving a rescue pack on hospital discharge is controversial as the hospital team is not, in general, the team that provides ongoing support to use these. There is thus recognised over- and under-use of rescue packs, associated harm from these medicines and variable provision. Providing a rescue pack, with education on how to use and support for when to use, has not been specifically tested in the high-risk 90-day period for readmission following a hospitalised exacerbation. It is the investigators' hypothesis that rescue packs on discharge in addition to a comprehensive self-supported management plan, consisting of the Asthma+Lung UK written management plan and twice weekly automated phone and or text messaging during this 90 day high risk period, will reduce readmissions by 20% compared to standard care.

Why is this research important in terms of improving the health of patients and health and care services?

Reducing re-admission through provision of supported rescue pack use would benefit people living with COPD and the NHS. A reduction in readmissions of 20% could save the NHS £86 million per quarter (£344 million per annum). Conversely, demonstrating that rescue packs are not effective when used in this way will address controversy about use, and reduce pressure on antimicrobial resistance and harm from over-use of oral corticosteroids. Integrated care systems are rapidly developing out-of-hospital support for people with exacerbations of COPD including digitally supported virtual wards. The proposed trial will define the role of supported rescue pack provision in the design and implementation of these programmes, enhancing their ability to reduce demands on urgent and acute care. Whether positive or negative, this trial will help to reduce the current variation in service provision by providing a definitive answer to the study question. Furthermore, preventing exacerbations of COPD have been identified as a priority by the James Lind Alliance (JLA) Priority Setting Partnership (PSP)12.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Individuals admitted to hospital with COPD exacerbation who have recently been discharged (discharged from ongoing support from secondary care team which includes hospital and virtual wards). Admission is defined as an episode in which a patient with an exacerbation of COPD is admitted to a ward and has stayed in hospital for 4 hours or more, including Emergency Medicine Centres, Medical Admission Units, Clinical Decision Units, short stay wards or similar but excludes patients treated transiently before being discharged from Emergency Department.
* Ability to provide written informed consent

Exclusion Criteria:

* Individuals who require invasive ventilation during the hospital admission
* Patients who have an expected survival of less than 90 days
* Patients with signs of new consolidation on chest X-ray (if available).
* Individuals who have been discharged to a residential or nursing home to residential or nursing home.
* Individuals who are unable to manage a supported self-management plan.
* Individuals with no access to telephone.
* Individuals who are already taking part in an interventional trial.
* Previous participation in the RAPID trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to first all-cause readmission within 90 days of discharge | Day 90
  Time to first all-cause readmission within 90 days of discharge.

SECONDARY OUTCOMES:
Time to and frequency of COPD-related readmissions at 30 days | Day 30
  Time to and frequency of COPD-related readmissions at 30 days post index discharge.
Time to and frequency of COPD-related readmissions at 90 days | Day 90
  Time to and frequency of COPD-related readmissions at 90 days post index discharge.
Days alive and out of hospital at day 90 | Day 90
  Days alive and out of hospital at day 90 post index discharge.
Time to and frequency of all COPD exacerbations at day 30 | Day 30
  Time to and frequency of all COPD exacerbations at day 30 post index discharge.
Time to and frequency of all COPD exacerbations at day 90 | Day 90
  Time to and frequency of all COPD exacerbations at day 90 post index discharge.
Cumulative systemic oral corticosteroids use over 90 days | Day 90
  Cumulative systemic oral corticosteroids use over 90 days post index discharge.
Cumulative systemic antibiotic use over 90 days | Day 90
  Cumulative systemic antibiotic use over 90 days post index discharge
Number of health care contacts at baseline, day 90 | Day 90
  Number of health care contacts at baseline, day 90 post index discharge
Number of health care contacts at baseline, day 180 | Day 180
  Number of health care contacts at baseline, day 180 post index discharge
Number of health care contacts at baseline and 1 year | Month 12
  Number of health care contacts at baseline, and 1 year post index discharge
All cause readmission at 30 days | 30 days
  All cause readmission at 30 days post index discharge
All cause-, cardiovascular- and COPD- related mortality at day 90 | Day 90
  All cause-, cardiovascular- and COPD- related mortality at day 90 post index discharge
All cause-, cardiovascular- and COPD- related mortality over 12 months | Month 12
  All cause-, cardiovascular- and COPD- related mortality over 12 months post index discharge
EQ-5D-5L Health questionnaire (quality of life) at 1 year | Month 12
  EQ-5D-5L Health Questionnaire score (quality of life) is used to ascertain participants' quality of life as reflected by their capacity for mobility, self care, usual activities, pain or discomfort, anxiety and depression. Mobility self care and usual activities components are graded from "no problems" to "unable to perform" (from best outcome to worst outcome respectively). Pain, anxiety and depression are graded on the scale from "none" to "extreme" (from best outcome to worst outcome respectively).
EQ-5D-5L Health questionnaire (quality of life) at day 90 | Day 90
  EQ-5D-5L Health Questionnaire score (quality of life) is used to ascertain participants' quality of life as reflected by their capacity for mobility, self care, usual activities, pain or discomfort, anxiety and depression. Mobility self care and usual activities components are graded from "no problems" to "unable to perform" (from best outcome to worst outcome respectively). Pain, anxiety and depression are graded on the scale from "none" to "extreme" (from best outcome to worst outcome respectively).
EQ-5D-5L Health questionnaire (quality of life) at day 180 | Day 180
  EQ-5D-5L Health Questionnaire score (quality of life) is used to ascertain participants' quality of life as reflected by their capacity for mobility, self care, usual activities, pain or discomfort, anxiety and depression. Mobility self care and usual activities components are graded from "no problems" to "unable to perform" (from best outcome to worst outcome respectively). Pain, anxiety and depression are graded on the scale from "none" to "extreme" (from best outcome to worst outcome respectively).
Incremental cost-effectiveness ratio (ICER, a ratio of the additional cost divided by the additional effectiveness of SRP compared to UC) at day 90 | Day 90
  Incremental cost-effectiveness ratio (ICER, a ratio of the additional cost divided by the additional effectiveness of SRP compared to UC) at day 90
Incremental cost-effectiveness ratio (ICER, a ratio of the additional cost divided by the additional effectiveness of SRP compared to UC) at day 180 | Day 180
  Incremental cost-effectiveness ratio (ICER, a ratio of the additional cost divided by the additional effectiveness of SRP compared to UC) at day 180
Incremental cost-effectiveness ratio (ICER, a ratio of the additional cost divided by the additional effectiveness of SRP compared to UC) at 1 year | Month 12
  Incremental cost-effectiveness ratio (ICER, a ratio of the additional cost divided by the additional effectiveness of SRP compared to UC) at 1 year
Qualitative interviews to examine and describe usual care | Day 90
  Interviews will be conducted by telephone, will take up to approximately 60 minutes, and will be audio-recorded using an encrypted device. They will follow a topic guide focusing on the participant's experience of the post-discharge intervention, including their knowledge of the use of rescue packs, whether they used a rescue pack and in what circumstances, their views on the support and guidance provided (written, telephone, and text message), and the fit of the intervention into their day-to-day lives.
Qualitative interview examination of fidelity to and adaptation of the plan in the intervention arm | Day 90
  Interviews will be conducted by telephone, will take up to approximately 60 minutes, and will be audio-recorded using an encrypted device. They will follow a topic guide focusing on the participant's experience of the post-discharge intervention, including their knowledge of the use of rescue packs, whether they used a rescue pack and in what circumstances, their views on the support and guidance provided (written, telephone, and text message), and the fit of the intervention into their day-to-day lives
Serious adverse events | Through study completion, average of 4 years
  Serious adverse events
Presence of bacterial resistance to antimicrobial agents | Through study completion, average of 4 years
  Proportion of isolates resistant to common antibiotics. This will be assessed via routine microbial laboratory antibiotic sensitivity
Quality of life COPD assessment Test (CAT) score at day 90 | Day 90
  Quality of life COPD assessment Test (CAT) score at day 90 post index discharge. The CAT is a validated, short (8-item) and simple patient completed questionnaire, with good discriminant properties, developed for use in routine clinical practice to measure the health status of patients with COPD. The CAT has a scoring range of 0-40, with 0 being the minimal score indicating no disease symptoms (better outcome) and 40 being the maximum indicating the greatest severity of COPD (worse outcome).
Quality of life COPD assessment Test (CAT) score at day 180 | Day 180
  Quality of life COPD assessment Test (CAT) score at day 180 post index discharge. The CAT is a validated, short (8-item) and simple patient completed questionnaire, with good discriminant properties, developed for use in routine clinical practice to measure the health status of patients with COPD. The CAT has a scoring range of 0-40, with 0 being the minimal score indicating no disease symptoms (better outcome) and 40 being the maximum indicating the greatest severity of COPD (worse outcome).
Quality of life COPD assessment Test (CAT) score at 1 year | Month 12
  Quality of life COPD assessment Test (CAT) score at 1 year post index discharge. The CAT is a validated, short (8-item) and simple patient completed questionnaire, with good discriminant properties, developed for use in routine clinical practice to measure the health status of patients with COPD. The CAT has a scoring range of 0-40, with 0 being the minimal score indicating no disease symptoms (better outcome) and 40 being the maximum indicating the greatest severity of COPD (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Mona Bafadhel, Professor, Principal Investigator — King's College London
Locations (34):
- United Kingdom (34):
  - Barnsley Hospital NHS Foundation Trust, Barnsley
  - University Hospitals Birminham NHS Foundation Trust, Birmingham
  - Blackpool Teaching Hospitals, Blackpool
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - University Hospitals Sussex NHS Foundation Trust, Brighton
  - North Bristol University Trust, Bristol
  - County Durham and Darlington NHS Foundation Trust, Durham
  - Gateshead NHS Foundation Trust, Gateshead
  - East Suffolk and North Essex Foundation Trust, Ipswich
  - University Hospitals of Morecambe Bay NHS Foundation Trust, Lancaster
  - University Hospitals of Leicester NHS Trust, Leicester
  - Cardiff and Vale University Health Board, Llandough
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - King's College Hospital, London
  - London North West University Healthcare NHS Trust, London
  - Royal Free London NHS Foundation Trust, London
  - Maidstone and Tunbridge Wells NHS Trust, Maidstone
  - South Tees NHS Foundation Trust, Middlesbrough
  - Milton Keynes University Hospital NHS Foundation Trust, Milton Keynes
  - Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Nottingham University Hospitals Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Rotherham NHS Foundation Trust, Rotherham
  - University Hospital Southampton NHS Foundation Trust, Shirley
  - Frimley Health NHS Foundation Trust, Slough
  - South Tyneside and Sunderland NHS Trust, South Shields
  - Southport and Formby District General Hospital, Southport
  - Stockport NHS Foundation Trust, Stockport
  - North Tees and Hartlepool NHS Foundation Trust, Stockton-on-Tees
  - Sherwood Forest Hospitals NHS Foundation Trust, Sutton in Ashfield
  - Somerset Foundation Trust, Taunton
  - Whiston Hospital, Whiston
  - Somerset Foundation Trust, Yeovil

IPD SHARING:
Plan to Share IPD: No
When the study is complete, a data sharing dataset will be created from the raw data by the study analyst, which will not include any other identifiable data and study PIN will be altered so that individuals are not recognisable from the dataset.
  The study will comply with the General Data Protection Regulations (GDPR).

DOCUMENTS (1):
  • Study Protocol (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT06347536/Prot_001.pdf